CLINICAL TRIAL: NCT00480922
Title: Randomized Controlled Trial Comparing the Effects of a Low Glycemic Load Diet With a Low Fat Diet on Hepatic Steatosis in Overweight Children and Adolescents
Brief Title: Effects of a Low Glycemic Load Diet on Fatty Liver in Children
Acronym: DELIVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-03-0092 (completed)
Record Dates: First submitted 2007-05-23; First posted 2007-05-31 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Hepatic Steatosis
Keywords: non-alcoholic fatty liver disease; steatohepatitis; overweight; insulin resistance
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease; Overweight; Insulin Resistance | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): A low glycemic load diet
  Interventions: Behavioral: Low glycemic load diet
- 2 (Active Comparator): Low fat diet
  Interventions: Behavioral: Low fat diet

INTERVENTIONS:
Behavioral: Low glycemic load diet — Outpatient behavioral counseling
  Arms: 1
Behavioral: Low fat diet — Outpatient behavioral counseling
  Arms: 2

SUMMARY:
There has been a recent increase in incidence of obesity and its associated morbidities, including T2 DM, hypertension and hepatic steatosis. Hepatic steatosis is a precursor to non-alcoholic steatohepatitis, cirrhosis and end-stage liver disease. The 1st reported case of pediatric hepatic steatosis was in 1980 and it is now affects 30-77% of overweight children. In addition to its association with obesity, hepatic steatosis has been associated with the metabolic syndrome, insulin resistance, and post-prandial hyperglycemia. Current treatment of hepatic steatosis includes weight loss with a hypocaloric low fat diet. Given the association with insulin resistance and post-prandial hyperglycemia, adult patients with hepatic steatosis that does not respond to weight loss are placed on insulin sensitizing drugs. We hypothesize that weight loss with a diet designed to decrease insulin resistance and post-prandial hyperglycemia, a low glycemic load diet, will provide a safe and effective way to decrease hepatic fat content in the pediatric population. This hypothesis will be tested with a randomized control trial comparing the effect of a low fat diet with a low glycemic load diet.

ELIGIBILITY:
Inclusion Criteria:

* BMI >95th percentile for age and sex
* Weight <300 pounds
* Ability to lie quietly in the MRI for approximately 45 minutes
* Willing and able to attend all sessions.
* Working telephone
* Greater than or equal to 10% hepatic steatosis on nMR spectroscopy

Exclusion Criteria:

* Any other medical condition besides obesity that may predispose to liver disease
* Medications that affect liver metabolism
* Any causes of chronic hepatitis
* Diabetes
* Inability to adhere to prescribed diets
* Currently on high-dose vitamins and not willing to discontinue
* Weight loss/gain in the past 6 months of >10% of total body weight.
* Sibling of any subject who is already enrolled
* Any alcohol consumption

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
percent liver fat as determined by nMR spectroscopy | 6 months

SECONDARY OUTCOMES:
hepatic steatosis as measured by T1 weighted MRI images | 6 monhts
visceral fat | 6 months
liver function tests | 6 months
measures of oxidative stress | 6 months
measures of chronic inflammation | 6 months
insulin resistance | 6 months
serum lipids | 6 months
blood pressure | 6 months
insulin secretion | baseline
measures of glucose tolerance | 6 months
adiponectin | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David S Ludwig, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Scribner KB, Pawlak DB, Ludwig DS. Hepatic steatosis and increased adiposity in mice consuming rapidly vs. slowly absorbed carbohydrate. Obesity (Silver Spring). 2007 Sep;15(9):2190-9. doi: 10.1038/oby.2007.260. PMID 17890486
- [Derived] Ramon-Krauel M, Salsberg SL, Ebbeling CB, Voss SD, Mulkern RV, Apura MM, Cooke EA, Sarao K, Jonas MM, Ludwig DS. A low-glycemic-load versus low-fat diet in the treatment of fatty liver in obese children. Child Obes. 2013 Jun;9(3):252-60. doi: 10.1089/chi.2013.0022. Epub 2013 May 24. PMID 23705885